CLINICAL TRIAL: NCT04138160
Title: Investigating the Effects of Two Weeks of 5:2 Intermittent Energy Restriction or Continuous Energy Restriction on Basal and Postprandial Metabolism in Normal-weight, Young Participants
Brief Title: Effects of Two Weeks of 5:2 Intermittent Energy Restriction on Basal and Postprandial Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 121-1809
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-10

CONDITIONS: Weight Loss
Keywords: obesity dietary restriction
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5:2 intermittent energy restriction (Experimental): The 5:2 intermittent energy restriction (IER) of 70% restriction (~600 kcal) delivered for two non-consecutive days/week and no restriction (so sufficient energy to meet the requirement of participants) on the other 5 days/week.
  Interventions: Other: 5:2 Intermittent energy restriction
- Continuous energy restriction (Other): The continuous energy restriction (CER) of 20% restriction below the estimated requirement of participants (~1600 kcal) 7 days/week.
  Interventions: Other: Continuous energy restriction

INTERVENTIONS:
Other: 5:2 Intermittent energy restriction — Substantial (70%) energy restriction for 2 non-consecutive days/week interspersed with normal energy intake (isoenergetic) on the remaining 5 days of the week.
  Other Names: 5:2 IER
  Arms: 5:2 intermittent energy restriction
Other: Continuous energy restriction — 20% energy restriction each day relative to the energy requirement.
  Other Names: CER
  Arms: Continuous energy restriction

SUMMARY:
Worldwide, a third of adults were overweight in 2016, and 13% were obese. Excess energy intake results in weight gain. Excess fat increases the risk of disease (eg. cardiovascular diseases, type 2 diabetes mellitus (T2DM), hypertension, dyslipidemia, dementia, certain cancers). Modest weight reduction (>5% of body weight) decreases the incidence and progression of many of these diseases. Daily energy restriction or continuous energy restriction (CER) involves diets that have a 500-600 kcal deficit per day resulting in sustainable weight loss. However, adherence is difficult. Diets following a 5:2 intermittent energy restriction (5:2 IER) pattern may be better. Approximately 75% energy restriction is maintained for 2 non-consecutive days/week and normal energy intake is consumed on the remaining 5 days of the week. Significantly reduced fasting insulin concentration and insulin resistance were shown in the 5:2 IER regimen compared with the CER regimen. In this study, normal-weight young participants will be recruited and 5:2 IER and CER will be compared over 2 week periods. Subcutaneous continuous glucose monitoring (CGM) devices will be undertaken. An ad libitum pasta meal will be consumed by participants three hours after the ingestion of breakfast to evaluate the energy intake. Postprandial thermogenesis in response to the test drink will be evaluated.

DETAILED DESCRIPTION:
Once participants have consented to be screened, they will come to the lab for a medical screening. If the medical screening is satisfactory, all participants will be asked to undergo a one-week pre-study standardization period. Participants will be asked to maintain their normal dietary and physical activity patterns throughout this period. Participants will be asked to complete a 3-day food diary, which will be analyzed to evaluate their habitual food intake and temporal distribution of energy intake throughout the day. In addition, participants will be provided with and instructed on how to use, an Actiheart (a device that combines accelerometry with heart rate monitoring). This device will be placed on the participants' chest using two standard electrocardiogram (ECG) electrodes to record HR, heart rate variability and activity level (to allow estimation of total energy expenditure) for one week. Both items will be returned before the next visit, which will be the pre-intervention measurement. After the pre-intervention visit, participants will be then randomly assigned to two weeks of either (1) the CER of 20% restriction below their estimated requirement (~1600 kcal) 7 days/week or (2) the 5:2 IER of 70% restriction (~600 kcal) delivered for two non-consecutive days/week and no restriction (so sufficient energy to meet their requirement) on the other 5 days/week. Seven days after the pre-intervention visit, participants will then start their 2-week intervention. A 7-day gap is designed in a bid to ensure both pre- and post-intervention measurements will be conducted during the second week of the follicular phase for females. The foods, drinks and overall energy restriction will be the same on each arm. Using estimated BMR based on the Henry equation and the individual daily physical activity level (PAL), estimated from the Actiheart during a one-week standardization period and the physical activity questionnaire, allowed the estimation of daily energy requirements for each subject using basal metabolic rate x PAL. Thus energy intake will be tailored to each participant's specific energy requirements. According to the suggestion from The Association of UK Dietitians, 2 non-consecutive ER days can be achieved on Day 1 and Day 4 of an IER week, thus the investigators will fix and prescribed the two ER days in a week with 3 days apart.

Food on intervention days will be prepared based on a 3-day sequence of menus to avoid boredom but be practical regarding the provision of foods. Each menu provides three meals/day to avoid confounding effects causing by altering meal frequency between the interventions. Three meals/day (and no snacks) is selected to make each eating incident acceptable on the most restricted day. Three meals with a macronutrient distribution of ~50% energy from carbohydrates, ~31% from fat and ~19% from protein will be prescribed. The distribution of energy across the day will be 25% of daily energy requirements from breakfast, 37.5% from lunch and 37.5% from the evening meal. To avoid confounding by altering the mealtime, and the period between which meals are consumed, breakfast will be instructed to be consumed between 8 am-8:30 am; lunch between 1 pm-1:30 pm and evening meal between 6 pm-6.30 pm. Menu designed so that it could be proportionally increased and decreased depending on the intervention requirement and informed by cooking facilities available and optimizing food safety. Participants will be instructed to adhere to the prescribed meal plan and record their food intake by taking photos.

On Day 7 of each experimental trial, participants will report to the unit in the morning after an overnight fast (~12h) for the assessment of body weight. The investigators will also use this visit to attach a subcutaneous continuous glucose monitoring (CGM) device, which will be placed on the abdomen to allow for the estimation of continuous blood glucose over the last 7 days of each trial. Also, the investigators will download the data from the pedometer and use it to assess compliance with the requirements of the study during the first week. CGM and pedometer will be removed upon arrival on the post-intervention visit.

On the day after one week pre-study standardization period and the day after the 2-week intervention, the participants will be asked to attend the laboratory after an overnight fast to undergo a series of appetite and metabolic measurements in response to a standardised breakfast in the form of a milk-based test drink (in a volume of 10 kcal/kg body weight and energy distribution from the macronutrients will be 47.9 % carbohydrate, 35.1% fat, and 17% protein) and a subsequent ad libitum pasta lunch containing cheese, olive oil, and tomato sauce, which will provide 148.24 kcal/100g with 49.8%, 15.4% and 34.8% energy provided by carbohydrates, protein and fat, respectively.

ELIGIBILITY:
Inclusion Criteria:

* ages between 20 - 35 years;
* healthy with a body mass index (BMI) between 20 and 27 kg·m-2;
* a waist circumference < 94 cm for males and < 80 cm for females;
* ability to give informed consent

Exclusion Criteria:

* smoking (including vaping);
* regularly skipping breakfast;
* any metabolic (e.g. diabetes), endocrine (e.g. hyperthyroidism) or cardiovascular (e.g. heart or blood) abnormalities including hypertension or heart failure;
* clinically significant abnormalities on screening including ECG abnormalities;
* taking routine medication that may alter cardiovascular function and blood flow (e.g. blood pressure-lowering drugs or drugs that cause hypertension);
* taking medication for diabetes or having diabetes;
* a history of substance abuse in the last six months;
* well-trained individuals with PAL>2.00;
* on an energy-restricted diet;
* high alcohol consumption (<3-4 units/d for men; <2-3 units/d for women);
* females who are pregnant or lactating and with irregular menstrual cycles;
* self-reported allergy, intolerance or strong dislike of foods or drinks to be offered for the test breakfast, pasta meal or during the intervention period;
* Beck Depression Inventory (BDI) score >10, and Eating Attitudes Test (EAT-26) score >20 as self-reported markers of symptoms and concerns characteristic of depression and eating disorders, respectively.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Incremental area under the curve for insulin | Over three hours from baseline
  Incremental area under the curve for serum insulin will be calculated using samples at 20 minute intervals between baseline and three hours.

SECONDARY OUTCOMES:
Incremental area under the curve for arterialised whole blood glucose | Over four hours post baseline
  Incremental area under the curve for arterialised whole blood glucose will be calculated using samples collected at 10 minute intervals between baseline and four hours.
Incremental area under the curve for composite appetite score | Over four hour from baseline
  Composite appetite score will be calculated using 100mm visual analogue score ratings of satiety, fullness, hunger and prospective food consumption collected very 20 minutes between baseline and four hours.
Weight of consumption of a pasta meal three hours after baseline | Three hours post baseline
  Weight of pasta consumed from a bowl refilled prior to being empty until participants feel comfortably full.
Incremental area under the curve for free fatty acid | Over three hours from baseline
  Incremental area under the curve for FFA will be calculated using samples at 20 minute intervals between baseline and three hours.
Incremental area under the curve for TAG | Over three hours from baseline
  Incremental area under the curve for TAG will be calculated using samples at 20 minute
Continuous glucose monitoring | Over last 6 days of intervention
  Average glucose of 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Ian Macdonald, PhD, Study Director — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Select State..., United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Only anonymised individual personal data will be shared, upon specific request from other researchers, for example, in order to undertake a meta analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When requested.
Access Criteria: On receipt of requests, data will be made accessible if agreed by both the University of Nottingham.